CLINICAL TRIAL: NCT06534580
Title: Developing and Refining a Virtual Reality Intervention That Will Help to Manage Pain for People Living With Advanced Cancer
Brief Title: Virtual Reality for Advanced Cancer Pain
Acronym: VRcan
Status: Active, not recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: Velindre NHS Trust (Other Government); Lancaster University (Other); Brighton and Sussex University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 158450
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Neoplasm Metastasis; Pain; Palliative Care
Keywords: virtual reality; Pain management
MeSH Terms: conditions — Neoplasm Metastasis; Pain; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Phase I: People living with advanced cancer and experiencing pain.
  Participants will complete two interviews. In each interview, they will use a Virtual Reality headset and discuss with the researcher the potential benefits, any changes they would make to the experiences, and how they might use it in practice.
  Interventions: Device: Virtual Reality
- Phase II: Participants: Staff working at participating sites, technology specialists, Patient and Public Involvement (PPI) representative.
  There will be a workshop at each participating site. Participants will work together to manualise the intervention so that it is ready for a feasibility trial and process evaluation.
  They will discuss the following:
  * Indications of use for virtual reality as a pain therapy
  * Frequency of use: recommended number of sessions, duration.
  * Barriers or facilitators that might impact the use of virtual reality.
  * Pain and other patient-reported outcomes identified.
  * What possible longer-term goals of using virtual reality as a pain therapy could include.
  * Guidance for specific settings, including safety considerations.
  * Operator instructions: patient or operator delivered.
  * Infection control management.
- Phase III: Participants: People living with advanced cancer and experiencing pain.
  During this phase, we will implement the recommendations from the manual from phase II. A headset will be available for use on an as needed basis at each study location. Participants will be asked to provide feedback each time they use the headset. Specific for data on pain, the Brief Pain Inventory (BPI) will be completed. This looks at pain severity as well as how much pain impacts their daily life. Whilst the availability of only one headset per site will limit the frequency of use, particularly for those who are outpatients, this is reflective of current availability of virtual reality headsets in each location. This data will generate recommendations for future research and clinical practice, including the consideration of the economic impact.
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — A range of virtual reality software, delivered through the "DR.VR" (TM) device.
  Groups: Phase I; Phase III

SUMMARY:
Background

Pain is commonly experienced by people who are living with advanced (incurable) cancer. There is evidence to suggest virtual reality could help to relieve this pain: however, this evidence is poor quality with the intervention poorly defined. A robustly co-designed intervention, with people who have advanced cancer and experience pain, will facilitate a better evidence-base.

Aim

To develop and refine a virtual reality intervention that will help people living with advanced cancer to manage pain.

Objectives

1. Explore and establish key components of a virtual reality intervention for people with advanced cancer in terms of effectiveness, acceptability and feasibility using in-depth interviews and focus groups with people living with advanced cancer and experiencing pain.
2. Develop and manualise a virtual reality intervention using co-design methodology.
3. User-test the intervention to refine further.

Methods

Multi-method design, incorporating multiple stakeholder perspectives, over three phases:

Phase I. Focus groups or individual interviews with a total of 40 people, from four locations (Brighton, Cardiff, Liverpool, & London), who have advanced cancer and experience pain.

They will use the virtual reality intervention and give feedback on what resonated with them and what they would change.

Phase II. Four focus groups (one at each study location) with multiple stakeholders. During this stage, the findings from phase 1 will be presented and a manual will be produced that gives guidelines on use of the virtual reality intervention.

Phase III. Up to 20 people living with advanced cancer and pain will user-test the intervention over an eight-week period. During this phase, the investigators will test if/how often the virtual reality is used as part of routine practice in each site and identify any barriers of use.

Anticipated Impact and Dissemination

1. A robustly co-designed intervention, ready for testing in a larger trial, to assess the clinical and cost effectiveness of virtual reality as a form of pain management.
2. Guidelines for the use of virtual reality in a clinical setting.

The results will be published through academic routes (peer-reviewed publications as well as presented at national and international conferences). The investigators will also work with our group of people with lived experience and an oversight committee to establish the best other routes to disseminate the findings to the public e.g., a social media campaign, leaflets to clinical settings, blog and vlog posts.

ELIGIBILITY:
Inclusion Criteria:

Patients will be considered eligible to participate if:

* Under the care of the specialist palliative care team or cancer centre
* A documented diagnosis of advanced cancer (Synonyms: "Palliative", "terminal", "incurable", "treatable but not curable") in their medical notes, confirmed by the clinical team.
* Adult (aged 18 years or over)
* Pain score in the last 7 days of ≥1 on Numerical Rating Scale [0-10]
* Full visual and auditory abilities
* No restriction in range of head and neck movement
* Capacity to consent to the study
* Fluent in English
* An estimated prognosis of longer than 6 months.

Professional/staff participants will be considered eligible if:

* a registered healthcare professional (doctors, nurses, allied health professionals, psychologists)
* employed by the study or location or by the virtual reality company.

Exclusion Criteria:

Patients will be excluded if:

* a diagnosis of epilepsy
* are imminently dying
* the clinical team feel it would be detrimental to participate
* do not meet the study inclusion criteria

Professional/staff participants will be excluded if:

• They are not employed by the study location, or the virtual reality company

We will document reasons for not participating, where offered.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From in- and out- patient hospital and hospice settings where people are under specialist palliative care services.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Data on the use of virtual reality for managing pain, from the perspective of people living with advanced cancer who experience pain. | 15 months
A pilot of the intervention, how it will be implemented, and how it is expected to work. | 15 months
A user-tested virtual reality intervention with a manual for use, including guidelines for use in clinical settings and research priorities | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicola White, PhD, Principal Investigator — University College, London; Ollie Minton, Principal Investigator — Brighton and Sussex University Hospitals NHS Trust
Locations (4):
- United Kingdom (4):
  - Brighton and Sussex University Hospitals NHS Trust, Brighton
  - Velindre University NHS Trust, Cardiff
  - Marie Curie Hospice, Liverpool, Liverpool
  - St Christophers Hospice, London, London

IPD SHARING:
Plan to Share IPD: Undecided